CLINICAL TRIAL: NCT06345612
Title: Impact of Eccentric Training Conducted in the Conditions of Normobaric Hypoxia, Normoxia and Creatine Supplementation on Metabolic Control, Muscle Strength Level, Maximum Oxygen Consumption (VO2max) in Patients With Type 1diabetes Mellitus
Brief Title: Impact of Eccentric Training in Hypoxia With Creatine on Metabolic Control and VO2max in Patients With Type 1 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Silesian Centre for Heart Diseases (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hypoxia-Exercise-DiabetesT1
Record Dates: First submitted 2024-02-23; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-02

CONDITIONS: Type 1 Diabetes
Keywords: exercise; eccentric exercise; hypoxia; type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity; Hypoxia | interventions — Creatine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1. exercise in hypoxia with creatine supplementation (Experimental): * training program in normobaric hypoxic chamber set to contain equivalent to an altitude of 2500 meters above sea level (indoor air composition: 15,4% of O2 and 84,7% of N)
  * with creatine supplementation
  Interventions: Behavioral: hypoxia; Dietary Supplement: creatine supplementation
- 2. exercise in hypoxia without creatine supplementation (Experimental): * training program in normobaric hypoxic chamber set to contain equivalent to an altitude of 2500 meters above sea level (indoor air composition: 15,4% of O2 and 84,7% of N)
  * without creatine supplementation
  Interventions: Behavioral: hypoxia; Dietary Supplement: no creatine supplementation
- 3. exercise in normoxia with creatine supplementation (Experimental): * the same training program in normoxic conditions
  * with creatine supplementation
  Interventions: Behavioral: normoxia; Dietary Supplement: creatine supplementation
- 4.exercise in normoxia without creatine supplementation (Experimental): * the same training program in normoxic conditions
  * without creatine supplementation
  Interventions: Behavioral: normoxia; Dietary Supplement: no creatine supplementation

INTERVENTIONS:
Behavioral: hypoxia — eccentric training program conducted within normobaric hypoxic chamber
  Arms: 1. exercise in hypoxia with creatine supplementation; 2. exercise in hypoxia without creatine supplementation
Behavioral: normoxia — eccentric training program conducted within normoxic conditions
  Arms: 3. exercise in normoxia with creatine supplementation; 4.exercise in normoxia without creatine supplementation
Dietary Supplement: creatine supplementation — 5g of creatine per day
  Arms: 1. exercise in hypoxia with creatine supplementation; 3. exercise in normoxia with creatine supplementation
Dietary Supplement: no creatine supplementation — no creatine supplementation
  Arms: 2. exercise in hypoxia without creatine supplementation; 4.exercise in normoxia without creatine supplementation

SUMMARY:
Exercise plays an important role in treatment of diabetes. In recent years exercise training in normobaric hypoxia is used in training programs for athletes and in rehabilitation and also commercially. The aim of the study is to assess the impact of eccentric training conducted in conditions of normobaric hypoxia or normoxia and creatine supplementation on metabolic control: profile and stability of glucose concentration, HbA1c value, hypoglycemia and insulin demand, as well as the level of muscle strength, VO2max and anthropometric parameters

DETAILED DESCRIPTION:
People with type 1 diabetes benefit from training in normobaric hypoxia - the composition of the air in the training room is: 15.4% oxygen 84.7% nitrogen, which corresponds to hypoxia at an altitude of 2,500 m above sea level. Hypoxia leads to the production of the hypoxia-inducible transcription factor HIF-1, which is a regulator of the expression of many genes responsible for angiogenesis, muscle hypertrophy and glucose stability.

Before starting the10 - week training program all participants will undergo preliminary examination by a cardiologist during which echocardiography and ECG will be conducted. Then the incremental exercise test and muscle strength test will be performed to determine aerobic capacity (VO2max) and select individual weights to train for each participant.

Patients enrolled to the study will be randomly assigned to one of the following 2 groups (training under normoxia or hypoxia conditions) and subgroups (with and without supplementation of creatine).

Randomization will be carried out in blocks of 4 people.

Training sessions will take place with the assistance of a personal trainer in the Hypoxia Laboratory and the Muscle Strength and Power Laboratory of Academy of Physical Education in Katowice twice a week for 60 minutes for a period of 10 weeks. The subjects will complete the same eccentric training program with individually selected weights.

Within whole training period glucose level will be monitored via Flash Glucose Monitoring system (Free Style Libre2). During training sessions concentration of asprosin, irisin, GH, IGF-1 within blood serum immediately before and afrer the first and last training will be assessed.

At baseline and after 10 weeks blood count, ALT, AST, creatinine, GFR, HbA1c, ACR (albumin/creatinine ratio) in a random urine sample, body weight, BMI, waist-hip circumference, body composition, quality of life according to the EQ-Worksheet questionnaire, daily insulin requirement, incremental exercise test, muscle strength test (1RM) will be investigated among all participants.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes of at least 10 years duration,
* low physical activity,
* BMI:20-31 kg/m2,
* treated with multiple insulin injections (at least 4 daily) or insulin pump (continuous subcutaneous insulin infusion [CSII]),
* negative ECG exercise test,
* HbA1c ≤ 8,0%,
* high knowledge about functional insulin therapy, carbohydrate counting and diabetes management during exercise,
* experience in use of FreeStyleLibre2 (Flash Glucose Monitoring System, Abbott),
* Informed consent to participate in research signed by enrolled subjects

Exclusion Criteria:

* HbA1c > 8,0%,
* advanced complications of diabetes [pre-proliferative or proliferative retinopathy, and previous laser therapy, microalbuminuria or overt nephropathy, autonomic neuropathy (including lack of elevated heart rate during physical activity)],
* patients physically active (regular physical activities more than once a week),
* positive ECG exercise test,
* history of cardiovascular event or coronary heart disease

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Metabolic control of diabetes | before and after 10 weeks
  HbA1c (%, mmol/mol)
Time in range | before and after 10 weeks
  TIR- percentage of time with blood glucose in a target range: 70-180 mg/dl (%)
Time below range | before and after 10 weeks
  TBR - percentage of time with blood glucose levels<70 mg/dl (%)
Maximum oxygen consumption (VO2max) | before and after 10 weeks
  measured during incremental exercise test

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Strojek, Prof., Study Chair — Medical University of Silesia in Katowice
Locations (1):
- Department of Internal Diseases, Diabetology and Cardiometabolic Disorders, School of Medicine with the Division of Dentistry in Zabrze, Medical University of Silesia in Katowice, Poland, Zabrze, Silesian Voivodeship, Poland